CLINICAL TRIAL: NCT00276458
Title: A Multicenter., Rand., Double-Blind, Titration Study to Evaluate & Compare the Efficacy & Safety of Ezetimibe Plus Atorvastatin Vs Atorvastatin in Hypercholesterolemic Pts. at Moderately High Risk for CHD Not Adequately Controlled on Atorvastatin 20 Mg
Brief Title: To Evaluate Ezetimibe Plus Atorvastatin Versus Atorvastatin in Patients With High Cholesterol Not Controlled on Atorvastatin 20 mg (0653-079)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-079; 2005_104
Record Dates: First submitted 2006-01-10; First posted 2006-01-13 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Atorvastatin 40mg tablet + Atorvastatin 20mg Pbo and ezetimibe 10mg Pbo tablets po qd (by mouth, once a day).
  Interventions: Drug: Comparator: atorvastatin; Drug: Comparator: Placebo
- 2 (Experimental): Atorvastatin 40mg Pbo tablet + Atorvastatin 20mg and ezetimibe 10mg tablets po qd (by mouth, once a day).
  Interventions: Drug: Comparator: ezetimibe; Drug: Comparator: Placebo.

INTERVENTIONS:
Drug: Comparator: atorvastatin — Atorvastatin 40mg tablet po qd (by mouth, once a day) for 6 weeks
  Arms: 1
Drug: Comparator: Placebo — Atorvastatin 20mg Pbo and ezetimibe 10mg Pbo tablets po qd (by mouth, once a day). for 6 weeks
  Arms: 1
Drug: Comparator: ezetimibe — Atorvastatin 20mg and ezetimibe 10mg tablets po qd (by mouth, once a day). for 6 weeks.
  Arms: 2
Drug: Comparator: Placebo. — Atorvastatin 40mg Pbo tablets po qd (by mouth, once a day). for 6 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate and compare the efficacy and safety of ezetimibe plus atorvastatin versus atorvastatin in hypercholesterolemic patients at moderately high risk for coronary heart disease not adequately controlled on atorvastatin 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patient with LDL-C >100 mg/dL & on a stable dose of atorvastatin 20 mg

Exclusion Criteria:

* Pregnant or lactating women or intending to become pregnant
* Patient with sensitivity or intolerance to ezetimibe or atorvastatin
* Patient with diabetes or coronary heart disease

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conard SE, Bays HE, Leiter LA, Bird SR, Rubino J, Lowe RS, Tomassini JE, Tershakovec AM. Efficacy and safety of ezetimibe added on to atorvastatin (20 mg) versus uptitration of atorvastatin (to 40 mg) in hypercholesterolemic patients at moderately high risk for coronary heart disease. Am J Cardiol. 2008 Dec 1;102(11):1489-94. doi: 10.1016/j.amjcard.2008.09.075. Epub 2008 Oct 23. PMID 19026302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In: 4/5/2006; Last Patient Last Visit 1/17/2008
  72 centers worldwide (US, Canada, Austria, Costa Rica)
  Eligible patients include those on a stable dose of atorvastatin 20 mg; or patients with adjusted LDL-C pre-screen ranges who were treated with other lipid modifying therapy, or were statin and/or ezetimibe naïve.
Pre-assignment Details: Patients received and were blinded to atorvastatin 20 mg for a 4/5- week run-in period.
  Patients needed an LDL-C ≥ 100 mg/dL and ≤ 160 mg/dL at Visit 2 (week -1). Eligible patients were randomized at Visit 3 (Week 0) to either atorvastatin 40 mg or addition of ezetimibe 10 mg to their 20 mg dose of atorvastatin for a 6-week treatment period.
Groups:
- Atorvastatin + Ezetimibe: Atorvastatin 20 mg + Ezetemibe 10 mg daily for 6 weeks
- Atorvastatin: Atorvastatin 40 mg Daily for 6 weeks
Period: Overall Study
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Started | 98 | 98
Completed | 92 | 91
Not Completed | 6 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Continuous [Mean (Full Range); unit: years] | 56.4 [24 to 78] | 58.0 [34 to 76] | 57.2 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 49 | 89
  Male | 58 | 49 | 107
Race/Ethnicity, Customized [Number; unit: participants]
  White | 58 | 60 | 118
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 8 | 15
  Black | 3 | 9 | 12
  Multi-Racial | 29 | 21 | 50
Apolipoprotein A-I [Mean (Standard Deviation); unit: mg/dL] | 161.8 (25.2) | 163.4 (24.6) | 162.6 (24.8)
Apolipoprotein A-I:Apolipoprotein B ratio [Mean (Standard Deviation); unit: Ratio] | 0.8 (0.2) | 0.7 (0.2) | 0.8 (0.2)
Apolipoprotein B [Mean (Standard Deviation); unit: mg/dL] | 122.9 (22.4) | 119.9 (21.0) | 121.4 (21.7)
C Reactive Protein [Mean (Standard Deviation); unit: mg/dL] | 1.6 (2.6) | 1.2 (1.7) | 1.5 (2.1)
High Density Lipoprotein (HDL) [Mean (Standard Deviation); unit: mg/dL] | 51.1 (12.1) | 51.7 (11.5) | 51.4 (11.8)
Low Density Lipoprotein (LDL) [Mean (Standard Deviation); unit: mg/dL] | 119.9 (19.4) | 117.9 (16.8) | 118.9 (18.1)
Low Density Lipoprotein Cholesterol (LDL-C):High Density Lipoprotein Cholesterol (HDL-C) ratio [Mean (Standard Deviation); unit: Ratio] | 2.4 (0.6) | 2.5 (0.7) | 2.4 (0.7)
Non- High Density Lipoprotein (Non-HDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 151.6 (24.1) | 148.4 (21.1) | 150.0 (22.7)
NonHigh Density Lipoprotein-Cholesterol (NonHDL-C):High Density Lipoprotein-Cholesterol (HDL-C)ratio [Mean (Standard Deviation); unit: Ratio] | 3.2 (1.0) | 3.0 (0.9) | 3.1 (1.0)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 202.6 (25.2) | 200.0 (21.5) | 201.3 (23.4)
Total cholesterol:High Density Lipoprotein Cholesterol (HDL-C) ratio [Mean (Standard Deviation); unit: Ratio] | 4.2 (1.0) | 4.0 (0.9) | 4.1 (1.0)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 152.5 (68.8) | 147.8 (75.3) | 149.0 (75.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C) at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 weeks
Population: Full Analysis Set (FAS): The FAS population includes all randomized patients who took at least 1 dose of study medication and had a baseline (BL) value and at least one post BL value. Post BL measurements up to 3 days following the last dose of double-blind study medication were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
Percent | -30.8 [-34.5 to -27.0] | -10.9 [-14.7 to -7.1]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline LDL-C value; Mean Difference (Final Values) = -19.9, 95% CI [-25.2 to -14.5], Standard Error of Mean 2.7 — (Atorva + EZ minus Atorva)

2. Secondary Outcome: Percent Change in High Density Lipoprotein -Cholesterol (HDL-C)at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
Percent | 3.2 [0.2 to 6.2] | 0.8 [-2.2 to 3.8]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p = 0.273, ANCOVA; Model terms: treatment and baseline HDL-C value; Mean Difference (Final Values) = 2.4, 95% CI [-1.9 to 6.6], Standard Error of Mean 2.1 — (Atorva + EZ minus Atorva)

3. Secondary Outcome: Percent Change in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
Percent | -26.7 [-30.1 to -23.3] | -10.2 [-13.6 to -6.9]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline non-HDL-C value; Mean Difference (Final Values) = -16.4, 95% CI [-21.2 to -11.7], Standard Error of Mean 2.4 — (Atorva + EZ minus Atorva)

4. Secondary Outcome: Percent Change From Baseline in Total-Cholesterol at Week 6
Description: ([6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
percent | -19.7 [-22.2 to -17.1] | -7.4 [-10.0 to -4.9]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline Total-C value; Mean Difference (Final Values) = -12.2, 95% CI [-15.8 to -8.6], Standard Error of Mean 1.8 — (Atorva + EZ minus Atorva)

5. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
Percent | -17.8 [-23.7 to -11.4] | -5.5 [-14.4 to 0.0]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p = 0.159, Nonparametric ANCOVA — ANCOVA using ranks based on normal scores (Tukey method) with model terms for treatment and baseline triglycerides value; ANCOVA using ranks based on normal scores (Tukey method) with model terms for treatment and baseline triglycerides value; Median Difference (Final Values) = -8.9, 95% CI [-17.7 to -0.4] — The median difference is based on the Hodges-Lehmann estimates of shift; The distribution-free 95% CI is based on Wilcoxon's rank sum test statistic. (Atorva + EZ minus Atorva)

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 89 | 90
Percent | -21.4 [-24.3 to -18.5] | -7.7 [-10.6 to -4.8]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline Apo B value; Mean Difference (Final Values) = -13.7, 95% CI [-17.8 to -9.6], Standard Error of Mean 2.1 — (Atorva + EZ minus Atorva)

7. Post Hoc Outcome: Percent Change in Apolipoprotein A-I at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 89 | 90
Percent | -1.9 [-4.2 to 0.4] | -1.2 [-3.5 to 1.1]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p = 0.681, ANCOVA; Model terms: treatment and baseline Apo A-I value; Mean Difference (Final Values) = -0.7, 95% CI [-3.9 to 2.6], Standard Error of Mean 1.6 — (Atorva + EZ minus Atorva)

8. Secondary Outcome: Percent Change From Baseline in Total-Cholesterol:High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
Percent | -20.6 [-23.7 to -17.5] | -7.5 [-10.6 to -4.4]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline Total-C:HDL-C value; Mean Difference (Final Values) = -13.1, 95% CI [-17.5 to -8.7], Standard Error of Mean 2.2 — (Atorva + EZ minus Atorva)

9. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C):High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
Percent | -31.9 [-35.8 to -27.9] | -11.0 [-14.9 to -7.0]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline LDL-C:HDL-C value; Mean Difference (Final Values) = -20.9, 95% CI [-26.5 to -15.3], Standard Error of Mean 2.8 — (Atorva + EZ minus Atorva)

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B: Apolipoprotein A-I Ratio at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 89 | 90
Percent | -19.0 [-22.3 to -15.6] | -5.8 [-9.2 to -2.5]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline Apo B:Apo A-I value; Mean Difference (Final Values) = -13.1, 95% CI [-17.9 to -8.3], Standard Error of Mean 2.4 — (Atorva + EZ minus Atorva)

11. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (HDL-C):High Density Lipoprotein Cholesterol (HDL-C) Ratio at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
Percent | -27.2 [-31.4 to -23.0] | -9.9 [-14.1 to -5.7]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline non-HDL-C:HDL-C value; Mean Difference (Final Values) = -17.3, 95% CI [-23.2 to -11.4], Standard Error of Mean 3.0 — (Atorva + EZ minus Atorva)

12. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein (CRP) at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 89 | 89
percent | -6.7 [-23.7 to 14.2] | -9.2 [-25.8 to 11.1]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p = 0.841, Longitudinal Data Analysis (LDA); LDA method of Liang and Zeger with model terms: treatment, time, and the interaction of time by treatment; Mean Difference (Final Values) = 2.5, 95% CI [-23.8 to 28.8] — Data for analysis was transformed by the natural log and the difference in geometric mean % change from BL calculated based on the difference in the back-transformed least squares means. (Atorva + EZ minus Atorva)

13. Post Hoc Outcome: Percent Change in C-Reactive Protein (CRP) at Week 6
Description: [(6 week value - baseline value)/baseline value]*100%.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 89 | 89
Percent | -19.2 [-25.0 to -4.0] | -9.1 [-22.2 to 5.3]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p = 0.839, Nonparametric ANCOVA; ANCOVA using ranks based on normal scores (Tukey method) with model terms for treatment and baseline CRP value; Mean Difference (Final Values) = -8.3, 95% CI [-26.1 to 8.3] — [estimate comment as in outcome 5, analysis 1]

14. Secondary Outcome: Number of Participants Who Attained Target LDL-C <100 mg/dL at Week 6
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Number analyzed (Participants) | 92 | 92
Participants
  <100 mg/dL | 77 | 45
  ≥100 mg/dL | 15 | 47
Statistical Analysis 1: Comparison: Atorvastatin + Ezetimibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Model terms: treatment and baseline LDL-C value; Odds Ratio (OR) = 8.60, 95% CI [3.80 to 19.47] — Estimated ratio is the predictive odds of attaining LDL-C target on Atorva + EZ versus Atorva

ADVERSE EVENTS:
Arm/Group | Atorvastatin + Ezetimibe | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/98
Other Adverse Events (participants affected / at risk) | 17/96 | 22/98
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin + Ezetimibe (N=96) | Atorvastatin (N=98)
Vertigo (Ear and labyrinth disorders) | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Chest Discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Edema (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (General disorders) | 1 | 1
Aspartate aminotransferase increased (General disorders) | 1 | 0
Blood creatinine phosphokinase increased (General disorders) | 0 | 1
Gamma-glutamyltransferase increased (General disorders) | 1 | 0
Transaminases increased (General disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
194 out of 196 randomized patients took at least one dose of blinded study therapy and were included in the safety analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.